CLINICAL TRIAL: NCT00801892
Title: OSA, Sleepiness, and Activity in Diabetes Management
Brief Title: Obstructive Sleep Apnea (OSA), Sleepiness, and Activity in Diabetes Management
Acronym: OSA_DM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eileen R. Chasens (Other)
Responsible Party: Sponsor-Investigator, Eileen R. Chasens, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: R21HL089522-01A2 (NIH)
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Results first posted 2014-03-27 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Sleep Apnea, Obstructive; Diabetes Mellitus, Type 2
Keywords: daytime sleepiness; obstructive sleep apnea; type 2 diabetes mellitus; diabetes management
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetes Mellitus, Type 2; Disorders of Excessive Somnolence | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Participants on sham-CPAP were allowed to try actual CPAP.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The mask and equipment appeared similar to actual CPAP but does not give pressure required to prevent OSA. Only CPAP naive persons eligible.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 subjects treated with CPAP (Active Comparator): Continuous Positive Airway Pressure treatment (CPAP)
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)
- 2 subjects treated with sham-CPAP (Sham Comparator): Sham Continuous Positive Airway Pressure treatment (sham-CPAP)
  Interventions: Device: Sham- Continuous Positive Airway Pressure (Sham-CPAP)

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — Mask worn over nose to splint open the airway with positive pressure to prevent the subject from holding their breath (apneas).
  Arms: 1 subjects treated with CPAP
Device: Sham- Continuous Positive Airway Pressure (Sham-CPAP) — Mask worn over nose to splint open the airway with positive pressure to prevent the subject from holding their breath (apneas).
  Arms: 2 subjects treated with sham-CPAP

SUMMARY:
Daily physical activity is important to achieve glucose control in persons with type 2 diabetes. The purpose of this study is to explore if obstructive sleep apnea and its daytime symptom, excessive sleepiness, act as barriers to physical activity. We will examine if treatment of obstructive sleep apnea with continuous positive airway pressure results in increased physical activity in persons with type 2 diabetes.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a serious disorder characterized by episodic obstruction of the pharyngeal airway accompanied by cessation or reduction in airflow. Untreated OSA has a negative impact 24 hours a day, disrupting nighttime sleep and causing excessive daytime sleepiness that interferes with functioning. Recent studies suggest that OSA and type 2 diabetes (T2DM) not only co-exist but that OSA may adversely affect glucose homeostasis. While physical activity is recognized as beneficial to persons with T2DM, OSA severity or daytime sleepiness may act to hinder persons with T2DM from participating in physical activity. The primary aim of this pilot/feasibility study is to obtain preliminary data to facilitate further hypothesis development and enhance the feasibility of conducting a double blind, randomized, placebo-controlled study to examine physical activity in subjects with T2DM and OSA who are treated with CPAP compared to subjects on sham-CPAP. The secondary aims are to explore: 1) the interrelationships of OSA severity, daytime sleepiness, and physical activity on glucose variability at baseline; 2) average pre-post therapy changes in glucose variability in subjects treated with CPAP compared to subjects receiving sham-CPAP, and 3) pre to post therapy changes in weight, diet, residual sleepiness and mood in subjects treated with CPAP compared to subjects receiving sham-CPAP.

The primary endpoint of the study, physical activity, will be measured by the Bodymedia SenseWear Pro Armband® to determine activity counts. The endpoint for glucose variability will be measured by the Medtronic Continuous Glucose Monitoring System (CGMS). Adherence to CPAP will be measured by a Smart Card® inserted in subjects' CPAP machines. We will limit the sample of subjects who are randomized to CPAP or sham-CPAP to persons with an adequate sleep duration pre-treatment (> 6 hours), with moderate or severe OSA and with EDS to have a more homogenous, profoundly affected sample for this pilot study. The information that will result from the proposed study on of the effect of OSA and EDS on glucose variability has the potential to lead to the development of improved behavioral interventions in persons with diabetes. In addition, this study contains measures of diet and mood to begin to elucidate the possible effects of OSA and EDS on diabetes management.

ELIGIBILITY:
Inclusion Criteria:

* T2DM (verified by primary care provider (PCP) or medication for T2DM)
* AHI (from PSG) greater than > 15
* A1c < 9.0%
* Epworth Sleepiness Sca;e > 10 (Baseline Assessment)
* Able to ambulate independently or with a cane
* Age 40-65 years
* BMI< 45
* No acute medical and psychiatric illness in past 3 months
* Self-reported sleep duration of at least 6 hours
* No changes in medications, including diabetic medications, in last 3 months
* Telephone access
* Able to perform study tests (e.g., speak, read and write in English)
* Willing to be randomized to CPAP or sham-CPAP

Exclusion Criteria:

* Diagnosis of another sleep disorder, in addition to OSA,
* Oxygen or Bi-level positive airway pressure required for treatment of OSA
* An oxygen saturation <75% for >10% of the diagnostic PSG or if subject has oxygen saturation <75% for >25% of the first 4 h of the diagnostic PSG
* Any individual in the household currently or with history of CPAP treatment
* Type 1 or gestational diabetes
* Prescribed insulin for treatment of type 2 diabetes
* Regular use (> 3 times/week) of hypnotic or alerting medications
* History of a near-miss or automobile accident due to sleepiness
* Employed in transportation-related safety sensitive occupation such as an airline pilot, truck driver, or train engineer
* Currently working night or rotating shifts
* Routine consumption of alcohol as determined by >2 drinks day
* Known allergy to medical adhesives or dermatological conditions that would preclude wearing CGMS
* Swim or water aerobics >once a week
* Participation in contact sports or activity that may damage CGMS device or cause injury from monitor
* Claustrophobia that prevents wearing the CPAP mask
* Pregnancy

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eileen R. Chasens, DSN, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1=Subjects With T2DM and OSA Who Are Treated With CPAP: subjects with T2DM and OSA who are treated with CPAP
  Continuous Positive Airway Pressure (CPAP): Worn over nose to splint open the airway and prevent the subject from holding their breath (apneas).
- 2=Sham-CPAP Then Active CPAP: subjects with T2DM and OSA who are treated with sham-CPAP originally; they were then allowed to cross over to the active CPAP after the main period
  Sham- Continuous Positive Airway Pressure (Sham-CPAP): Worn over nose to splint open the airway and prevent the subject from holding their breath (apneas).
Period: Main Study Period
Arm/Group | 1=Subjects With T2DM and OSA Who Are Treated With CPAP | 2=Sham-CPAP Then Active CPAP
Started | 12 | 11
Completed | 12 | 10
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Sham Crossover Period
Arm/Group | 1=Subjects With T2DM and OSA Who Are Treated With CPAP | 2=Sham-CPAP Then Active CPAP
Started | 0 | 7
Completed | 0 | 5
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: Sample primarily middle aged adults with type 2 diabetes
Groups:
- 2=Subjects With T2DM and OSA Who Are Treated With Sham-CPAP: subjects with T2DM and OSA who are treated with sham-CPAP
  Sham- Continuous Positive Airway Pressure (Sham-CPAP): Worn over nose to splint open the airway and prevent the subject from holding their breath (apneas).
- Total: Total of all reporting groups
Arm/Group | 1=Subjects With T2DM and OSA Who Are Treated With CPAP | 2=Subjects With T2DM and OSA Who Are Treated With Sham-CPAP | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.58 (10.98) | 53.45 (10.33) | 55.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23
BMI [Mean (Standard Deviation); unit: kg/m2] | 36.2 (6.9) | 34.8 (5.6) | 35.5 (6.2)
Education [Mean (Standard Deviation); unit: years] | 13.9 (3.5) | 14.4 (2.9) | 14.1 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity, Steps Walked
Description: Steps walked measured by the Bodymedia SenseWear Pro Armband®Data collected from the main study period
Time Frame: after one-month treatment
Measure: Mean (Standard Deviation); unit: steps walked
Arm/Group | 1=Subjects With T2DM and OSA Who Are Treated With CPAP | 2=Subjects With T2DM and OSA Who Are Treated With Sham-CPAP
Number analyzed (Participants) | 12 | 11
steps walked
  Baseline | 5892 (3841) | 6071 (2714)
  After one month | 6284 (3480) | 6684 (2509)

2. Secondary Outcome: Fructosamine
Description: Change in fructosamine level from baseline to one month: data from main study period
Time Frame: after one-month
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | 1 Subjects Treated With CPAP | 2 Subjects Treated With Sham-CPAP
Number analyzed (Participants) | 12 | 10
umol/L
  Baseline | 261 (37) | 267 (44)
  One Month | 253 (42) | 270 (48)

3. Secondary Outcome: Change in Sleep Quality
Description: From Pittsburgh Sleep Quality Index; scores range from 0 to 21 with higher scores worse sleep quality; data from main study period
Time Frame: after one month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 Subjects Treated With CPAP | 2 Subjects Treated With Sham-CPAP
Number analyzed (Participants) | 12 | 11
units on a scale
  Baseline | 10.33 (3.12) | 10.44 (5.29)
  One Month | 7.63 (3.96) | 9.78 (3.70)

4. Secondary Outcome: Change in Daytime Sleepiness During Main Study Period
Description: Daytime Sleepiness measured by the Epworth Sleepiness Scale; measured from 0 to 24; higher scores indicate worse sleepiness
Time Frame: after one month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 Subjects Treated With CPAP | 2 Subjects Treated With Sham-CPAP
Number analyzed (Participants) | 12 | 11
units on a scale
  Baseline | 11.42 (4.6) | 10.55 (3.7)
  After one month | 9.08 (5.7) | 10.50 (3.6)

5. Secondary Outcome: Change in Vigor-Activity During Main Study Period
Description: Vigor-Activity from Profiles of Mood Scale; scores range from 0 to 32 with higher scores indicating higher vigor/activity
Time Frame: after one month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 Subjects Treated With CPAP | 2 Subjects Treated With Sham-CPAP
Number analyzed (Participants) | 12 | 11
units on a scale
  Baseline | 15.08 (5.16) | 17.45 (7.02)
  One Month | 16.75 (6.63) | 10.70 (5.23)

6. Secondary Outcome: Fatigue/Inertia
Description: Fatigue/Inertia from the Profile of Moods Subscale; scores range from 0 to 28; higher scores indicate more fatigue/inertia
Time Frame: after one month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 Subjects Treated With CPAP | 2 Subjects Treated With Sham-CPAP
Number analyzed (Participants) | 12 | 11
units on a scale
  Baseline | 11.75 (4.3) | 9.36 (6.04)
  One Month | 9.08 (6.19) | 10.70 (5.23)

ADVERSE EVENTS:
Groups:
- 1 Subjects With T2DM and OSA Who Are Treated With CPAP: subjects with T2DM and OSA who are treated with CPAP
  Continuous Positive Airway Pressure (CPAP): Worn over nose to splint open the airway and prevent the subject from holding their breath (apneas).
- 2 = Subjects With T2DM and OSA Who Are Treated With Sham-CPAP: subjects with T2DM and OSA who are treated with sham-CPAP
  Sham- Continuous Positive Airway Pressure (Sham-CPAP): Worn over nose to splint open the airway and prevent the subject from holding their breath (apneas).
Arm/Group | 1 Subjects With T2DM and OSA Who Are Treated With CPAP | 2 = Subjects With T2DM and OSA Who Are Treated With Sham-CPAP
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes